CLINICAL TRIAL: NCT06438263
Title: An Open-label, Phase 1, Single Dose, Randomized, Parallel-group Study to Assess the Relative Bioavailability of Rocatinlimab (AMG 451) Autoinjector and Vial in Healthy Subjects
Brief Title: A Study to Evaluate Bioavailability of Rocatinlimab Autoinjector and Vial in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220014
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Rocatinlimab; AMG 451; Dermatology; Pharmacokinetics; Safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will be randomized to receive a single dose of rocatinlimab vial solution for SC injection.
  Interventions: Drug: Rocatinlimab
- Treatment B (Experimental): Participants will be randomized to receive a single dose of rocatinlimab autoinjector for SC injection.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Vial supplied as a single-use preservative free solution for SC injection.
  Other Names: AMG 451
  Arms: Treatment A
Drug: Rocatinlimab — Autoinjector for SC injection.
  Other Names: AMG 451
  Arms: Treatment B

SUMMARY:
The main objective of this study is to evaluate the pharmacokinetics (PK) of rocatinlimab given as a single subcutaneous (SC) autoinjector dose compared to vial in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent before initiation of any study-specific activities/procedures.
2. Healthy male or female participants, between 18 and 60 years of age (inclusive)
3. Body mass index between 18 and 32 kg/m2 (inclusive)

Exclusion Criteria:

1. History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
2. History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Check-in.
3. A QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 msec in male participants or > 470 msec in female participants or history/evidence of long QT syndrome at Screening or Check-in.
4. Systolic blood pressure ≥ 140 mmHg or ≤ 90 mmHg, or diastolic blood pressure ≥ 90 mmHg or ≤ 50 mmHg, or pulse rate ≥ 100 bpm or ≤ 40 bpm
5. History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee). Participants with seasonal allergies will be permitted.
6. Estimated glomerular filtration rate less than 70 mL/min/1.73 m2
7. Alanine aminotransferase or aspartate aminotransferase > 1.5 times the upper limit of normal at Screening or Check-in.
8. Positive hepatitis B or hepatitis C panel (including positive hepatitis B surface antigen [HBsAg] and/or positive hepatitis C antibody) and/or positive human immunodeficiency virus test at Screening. Participants whose results are compatible with prior hepatitis B vaccination (positive hepatitis B surface antibody, negative hepatitis B core antibody, negative HBsAg) or prior infection (positive hepatitis B core antibody, positive hepatitis B surface antibody, negative HBsAg) may be included.
9. Participants who have received live vaccines within 5 weeks prior to Screening, or plan to receive live vaccines within 90 days after administration of an investigational product.

   Inactive vaccination (e.g., non-live or nonreplicating agent), including coronavirus-2019 (COVID-19) vaccination, is allowed.
10. History of latent tuberculosis or active chronic, recurrent, or acute infection requiring treatment with systemic antibiotics, antiviral, antiparasitic, antiprotozoal, or antifungals which has not completely resolved, or for which therapy has not been completed, within 4 weeks before Screening.
11. Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before Check-in, excluding the following:

    1. Acetaminophen (paracetamol) (up to 2 g per day) for analgesia will be allowed.
    2. Hormonal contraception listed in Appendix 3 will be allowed.
    3. Hormone replacement therapy (e.g., estrogen) and hormonal contraceptives will be allowed.
12. All herbal medicines (e.g., St. John's wort), vitamins, and supplements consumed by the participant within the 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee) and in consultation with the Sponsor.
13. Participant has received a dose of an investigational drug within the past 90 days or 5 half-lives, whichever is longer, prior to Check-in.
14. Have previously completed or withdrawn from this study or any other study investigating rocatinlimab or have previously received rocatinlimab.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Rocatinlimab | Up to approximately 112 days
Area Under the Serum Concentration-time Curve (AUC) From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Rocatinlimab | Up to approximately 112 days
AUC From Time Zero to Infinity (AUCinf) of Rocatinlimab | Up to approximately 112 days

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Approximately 20 weeks
  TEAEs are any adverse events (AEs) that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms (ECG), and clinical laboratory tests that occurred after study treatment administration will be recorded as TEAEs.
  A serious AE (SAE) is defined as any AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgment may jeopardize the participant or may require medical or surgical intervention to prevent any of the outcomes listed above.
Number of Participants with Anti-rocatinlimab Antibodies | Up to approximately Day 112

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Fortrea Clinical Research Unit - Daytona Beach, Daytona Beach, Florida
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas
  - Fortrea Clinical Research Unit Inc. - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com